CLINICAL TRIAL: NCT00484549
Title: National, Multicenter, Prospective Study of Screening of Fabry Disease in a Population of Men Over 28 Days Old and Less Than 55 Years, Hospitalized for an Ischemic Stroke.
Brief Title: Fabry : National Initiative of Screening
Acronym: FIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Pierre CLAVELOU, CHU Clermont-Ferrand
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CHU63-0019
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2009-12-21 (Estimated); Status verified 2009-12

CONDITIONS: Ischemic Stroke Hospitalized
Keywords: Fabry disease, Screening, Ischemic stroke
MeSH Terms: conditions — Fabry Disease; Ischemic Stroke | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Procedure: Blood sample — Ischemic stroke hospitalized

SUMMARY:
Fabry disease is a genetic disease due to an enzymatic deficit. A screening of this disease allows patients to benefit from an enzyme replacement therapy and prevent the occurrence of life threatening manifestations such as an ischemic stroke.

The purpose of the study is to determinate the prevalence of Fabry disease in a population of male patients hospitalized for an ischemic stroke.

This study, with a screening of Fabry disease, allows the patients to make a precise diagnosis of their ischemic stroke and to facilitate the screening of the other members at the facility.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized ischemic stroke
* Written and signed informed consent from patient or legal representative

Exclusion Criteria:

* Patients belonging to a family which has a Fabry disease's diagnosis confirmed

Ages: 28 Days to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 889 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Fabry disease's screening (Positive microdosage confirmed by a macrodosage) | Positive microdosage confirmed by a macrodosage

SECONDARY OUTCOMES:
Describe and compare the characteristics of patients affected by Fabry disease and patients who are not affected Identify clinical and neuroradiological predictive elements of Fabry disease | patients affected by Fabry disease

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Clavelou, Pr, Principal Investigator — Unaffilliated
Locations (1):
- Hôpital Gabriel Montpied, Clermont-Ferrand, France

REFERENCES:
- [Background] Clavelou P, Besson G, Elziere C, Ferrier A, Pinard JM, Hermier M, Artigou JY, Germain DP. [Neurological aspects of Fabry's disease]. Rev Neurol (Paris). 2006 May;162(5):569-80. doi: 10.1016/s0035-3787(06)75051-2. French. PMID 16710123